CLINICAL TRIAL: NCT01621334
Title: Stage 1B Study Motivating Substance Abusing Batterers to Seek Treatment.
Brief Title: The Men's Domestic Abuse Check-Up Engages Adult Men Concerned About Their Abusive Behavior and Alcohol or Drug Use
Acronym: MDACU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lyungai Mbilinyi, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37863-C; R01DA017873 (NIH)
Record Dates: First submitted 2011-08-16; First posted 2012-06-18 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Domestic Violence; Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Enhancement Therapy (Experimental): Motivational Enhancement Therapy
  Interventions: Behavioral: Motivational Enhancement Therapy
- Educational brochure (Other): Intimate Partner Violence, Substance Abuse, and HIV risky behaviors Education
  Interventions: Behavioral: Educational information

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy — Two personal feedback sessions with counselor using motivational interviewing strategies.
  Arms: Motivational Enhancement Therapy
Behavioral: Educational information — Educational brochure about legal, health and behavioral effects of intimate partner violence, substance abuse, and HIV risky behaviors
  Arms: Educational brochure

SUMMARY:
This research is a stage 1b developmental trial evaluating an intervention called "The Men's Domestic Abuse Check-Up" with adult men abusing their intimate partners and also struggling with alcohol or drug use.

DETAILED DESCRIPTION:
One hundred and forty adult men concerned about their substance use and behaviors toward intimate partners, recruited in Washington State, will be enrolled in the trial. Participants are recruited through print and radio ads. Following a baseline assessment, participants are then randomly assigned to receive one of two interventions:

* The experimental intervention is a two-session motivational enhancement treatment. A personalized feedback report, containing information from the participant's assessment as well as normative comparison data, is reviewed, with the counselor employing motivational interviewing strategies intended to impact study outcomes.
* The comparison condition involves an educational brochure focusing on the legal, health and behavioral effects of intimate partner violence, substance abuse, and HIV risky behaviors.

Following the two interventions, participants are reassessed at 1 week, 1 month, and 4 months following either intervention.

ELIGIBILITY:
Inclusion Criteria:

* age (18 years and older)
* gender (male)
* self-reported abusive behaviors
* concerned about alcohol or drug use

Exclusion Criteria:

* not fluent in English
* they have a thought disorder that precludes full participation
* they refuse to accept randomization to condition

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
treatment seeking | 4 months

SECONDARY OUTCOMES:
self-report of intimate partner violence and substance use | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Lyungai F Mbilinyi, PhD, Principal Investigator — University of Washington School of Social Work
Locations (1):
- Innovative Programs Research Group, School of Social Work, University of Washington, Seattle, Washington, United States